CLINICAL TRIAL: NCT07103759
Title: Project REST: Club Sports
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID 2020 pandemic, unable to start recruitment.
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, MICHAEL A GRANDNER, Associate Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2002361146
Record Dates: First submitted 2020-02-10; First posted 2025-08-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Poor Quality Sleep
Keywords: Educational Intervention; Insomnia; Daytime Sleepiness; College Students; Athletes; Club Sports; Sleep Duration; Sleep Quality; Stress; Academic Stress
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Disorders of Excessive Somnolence

STUDY DESIGN:
Intervention Model Description: N=50 participants will be randomized to one of two groups.
  Group 1| N=25 participants will use the Project REST platform and also use one of the learned techniques. The applied technique they will be asked to complete will be to refrain from drinking caffeinated drinks late in the afternoon.
  Group 2|(N=25) will consist of participants using just the Project REST platform (control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project REST Platform+refrain from caffeine technique (Experimental): N =25 participants will use the Project REST platform and also use one of the learned techniques. The applied technique they will be asked to complete will be to refrain from drinking caffeinated drinks late in the afternoon.
  Interventions: Behavioral: Refrain from caffeine techniques; Behavioral: Project REST Platform
- Project REST Platform ONLY (Active Comparator): N =25 participants will consist of participants using just the Project REST platform (control group)
  Interventions: Behavioral: Project REST Platform

INTERVENTIONS:
Behavioral: Refrain from caffeine techniques — Participants will be asked to refrain from drinking caffeinated beverages in the late afternoon and evening.
  Arms: Project REST Platform+refrain from caffeine technique
Behavioral: Project REST Platform — Participants will use the Project REST platform

SUMMARY:
Evidence suggests that student athletes frequently experience sleep problems and are aware of the impact of sleep loss on mental and physical outcomes. As such, student athletes are motivated to improve sleep quality in order to improve their outcomes for overall athletic performance. This study will consist of two parts. The first part will be a survey given to 15 clubs early into the spring semester (this time will allow poor sleep habits and quality a chance to manifest). Of the individuals that participate, a survey will assess multiple domains of student athlete health, namely, sleep duration and quality, mood and depression, stress, and mental and physical well-being. The responses to the survey will be confidential, and at the end of the semester, students will be invited to complete the survey again Part 2 is an intervention. 50 of the participants will be chosen to partake in the intervention, based on predetermined criteria. The intervention will include an information session where students may ask questions. Students will be sent brief email reminders about adherence to the program and will be asked to monitor their sleep quality with sleep diaries. Half of the 50 chosen (25 students) will be asked to refrain from drinking caffeinated drinks (coffee, energy drinks, soft drinks, etc.) late in the afternoon (6pm and on). Caffeine can delay the bodies circadian rhythm and reduce the total sleep time.

DETAILED DESCRIPTION:
Over the past few years, the effects of a poor sleep in varsity level, collegiate student-athletes has been attributed to a broad range of physiologic, social, and environmental pressures, including long hours, additional stress, travel burden, and other sources. Studies have shown that chronic sleep deprivation and inadequate sleep are strongly associated with the development of cardiometabolic disease risk factors obesity, depression, anxiety disorders, alcohol use, other substance use, poorer academic performance, and reduced mental well-being, in addition to poorer athletic performance.

In data from student-athletes in the American College Health Association from 2011-2014, when asked about access to health-related information, sleep was one of the most infrequently-provided domains of information. Yet, more than half of the student-athletes reported that they wanted more information about sleep, more than nearly all other categories of information. In addition, sleep problems were common, such that 19.8% reported that sleep difficulties had been "traumatic or very difficult," 21.8% reported "extreme difficulty" falling asleep ≥3 nights/week, and 57.0% indicated that they got enough sleep to feel rested on ≤3 nights/week (20.4% ≤1 day/week). Regarding daytime consequences, 60.9% reported extreme tiredness ≥3 days/week and 17.7% reported that sleep difficulties interfered with academics. Additional data from this cohort shows that poor sleep was also associated with lower academic performance, worse mental health, increased substance use, and increased risky behaviors while drinking.

For this reason, we developed Project REST (Recovery Enhancement and Sleep Training) to be a program that can improve sleep among student athletes, despite the many situational constraints. The original Project REST study pilot study included educational, tracking, support, and motivational enhancement. This combination produced strong results, including 77 minutes increased sleep duration, 10% increased sleep efficiency, 55% improvement in sleep latency, 40% improvement in insomnia symptoms, 80% reduction in drowsy driving, and 21% improved overall energy level.

The University of Arizona has many men and women competing in Division 1 athletics in the public eye, but there are many other student athletes that also participate in sport. According to data collected from UA, there are 35 athletics organizations-- clubs that in most cases are not recognized by the National Collegiate Athletic Association (for example, rugby, lacrosse, etc.). With more than 1,000 UA student athletes competing regionally, nationally, and occasionally in cities around the world, the likelihood of similar poor sleep habits and diminished sleep quality are high. Using the platform of Project REST, the goal of this new study, Project REST: Club Sports, will be to inform, educate, and monitor a small pool of club sports student athletes and implementing the data collected into a program that can be dispersed to a larger audience.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate
2. Currently active on the team roster
3. Age 18 years or older

Exclusion Criteria:

1. Participant is under 18 years old
2. Not currently active on the team roster
3. Have medical conditions that the PI considers would preclude them from participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-24 (Estimated); Primary Completion 2021-02-24 (Estimated); Study Completion 2021-02-24 (Estimated)

PRIMARY OUTCOMES:
Changes in Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to post-intervention, around 6 weeks after baseline
  Change in Pittsburgh Sleep Quality Index (PSQI) score at the end of the 6-week intervention. The PSQI global score has a possible range of 0-21 points. A total score of 5 or above indicates overall poor sleep quality.
Changes in Insomnia Severity Index (ISI) | Change from baseline to post-intervention, around 6 weeks after baseline
  Change Insomnia Severity Index (ISI) score at the end of 6-week intervention. The Insomnia Severity Index is a frequently-used questionnaire to measure insomnia symptoms. Total score categories: 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Changes in Center for Disease Control (CDC) and Prevention Health-Related Quality of Life Scale (HRQOL) Score (Unhealthy Days) | Change from baseline to post-intervention, around 6 weeks after baseline
  Change in CDC Health-Related Quality of Life Scale (HRQOL) score at the end of 6-week intervention. Health-related quality of life (HRQOL) is an individual's or a group's perceived physical and mental health over time. Unhealthy days are an estimate of the overall number of days during the previous 30 days when the respondent felt that either his or her physical or mental health was not good. The minimum number of unhealthy days is 0 and the maximum is 30. A higher score means more unhealthy days, a worse outcome.
Changes in Center for Disease Control (CDC) and Prevention Health-Related Quality of Life Scale (HRQOL) Healthy Days | Change from baseline to post-intervention, around 6 weeks after baseline
  Change in healthy days from the CDC Health-Related Quality of Life Scale (HRQOL) at the end of 6-week intervention. Health-related quality of life (HRQOL) is an individual's or a group's perceived physical and mental health over time. Healthy days are the positive complementary form of unhealthy days.
  Healthy days estimates the number of recent days when a person's physical and mental health was good (or better) and is calculated by subtracting the number of unhealthy days from 30 days.The minimum number of healthy days is 0 and the maximum is 30. A higher number of healthy days is a better outcome.
Changes in Centers for Epidemiological Studies Depression (CESD) | Change from baseline to post-intervention, around 6 weeks after baseline
  Change in Centers for Epidemiological Studies Depression Scale (CESD) score at the end of 6-week intervention.
  Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Changes in Perceived Stress Scale (PSS) | Change from baseline to post-intervention, around 6 weeks after baseline
  Change in Perceived Stress Scale (PSS) score at the end of the 6-week intervention.The PSS is comprised of 14 items intended to measure how unpredictable, uncontrollable, and overloaded individuals find their life circumstances.Participants rate items on a 5-point Likert scale, ranging from 0 - "Never" to 4 - "Very often." Scores range from 0-56 higher scores indicate greater perceived stress.
Changes in Generalized Anxiety Disorder 7-item Scale (GAD-7) | Change from baseline to post-intervention, around 6 weeks after baseline
  Change in GAD-7 at the end of the 6-week intervention which is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. It contains 7 items with answers ranging from "Not at all" to "Nearly every day".

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Grandner, PhD, MTR, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States